CLINICAL TRIAL: NCT04697537
Title: Dexmedetomidine as Adjunct Medication to Local Infiltration Anesthesia (LIA) vs Ultrasound-Guided Regional Anesthesia (USRA) in Regard to Patients' Need for Opioids, Wellbeing, Satisfaction, and Knee Functionality in Knee-endoprosthetics
Brief Title: Ultrasound-guided Regional Anesthesia vs Local Infiltration Anesthesia With Dexmedetomidine and Ropivacaine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GAS1.0
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Pain, Postoperative; Anesthesia, Local; Gonarthrosis
MeSH Terms: conditions — Pain, Postoperative; Osteoarthritis, Knee | interventions — Dexmedetomidine; Ropivacaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided regional anesthesia (Active Comparator): Patient will be given a peripheral nerve block from their treating anesthesiologist before the operation (in the OR) with an conventional ultrasound guided femoral and sciatic block of each 15 ml ropivacaine 0,5% and 0,5 ml dexmedetomidine (100µg/ml).
  Interventions: Drug: Ultrasound guided regional anesthesia
- Local infiltration analgesia (Active Comparator): Patient will be given a local infiltration analgesia from their treating surgeon during the operation (in the OR) with 60 ml ropivacaine 0,5% and 1 ml dexmedetomidine (100µg/ml).
  Interventions: Drug: Local infiltration analgesia

INTERVENTIONS:
Drug: Ultrasound guided regional anesthesia — Applied perineurally preoperatively ultrasound guided regional anesthesia
  Other Names: dexmedetomidine; Ropivacaine
  Arms: Ultrasound guided regional anesthesia
Drug: Local infiltration analgesia — Applied in the wound intraoperatively from the orthopedics
  Other Names: dexmedetomidine; Ropivacaine
  Arms: Local infiltration analgesia

SUMMARY:
Evaluation of the Impact of dexmedetomidine as an adjunct for local infiltrations analgesia and ultrasound-based regional anaesthesia as pain medication in regard to patients' opioid need the first 48 hours after the total knee replacement operation.

DETAILED DESCRIPTION:
Evaluation of the Impact of dexmedetomidine as an adjunct for local infiltrations analgesia and ultrasound-based regional anaesthesia as pain medication in regard to patients' opioid need the first 48 hours after the total knee replacement operation. Secondary objectives are: Pain assesment, Pain medication necessary, functionality of the prothesis, satisfaction, wellbeing, postoperative discomforts, complications (delirium, allergic reactions, cardiopulmonary decompensation), procedure specific time.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* non pregnant
* patients with gonarthrosis who have given written consent for participation

Exclusion Criteria:

* Age below 18 years
* pregnancy
* breast-feeding patients
* allergies against study medication
* missing or denied written consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Need of opioid consumption in oral morphine equivalent | 48 hours postoperatively
  consumed opioids in mg of oral morphine equivalent

SECONDARY OUTCOMES:
Pain assesment | 5 days postoperatively or until discharge
  Pain experienced by patients according to self-assesment according to NRS (Numeric rating scale) (minimum 0, maximum 10) (higher score means worse outcome)
Pain medication necessary | 5 days postoperatively or until discharge
  Need of opioid consumption in mg of oral morphine equivalent up to the 5th postoperative day
Functionality of the prothesis - OKS (Oxford Knee Score) | 5 days postoperatively or until discharge
  According to physical examination by the Oxford Knee Score (minimum 0, maximum 48) (higher score means better outcome)
Functionality of the prothesis- KOOS (Knee Injury and Osteoarthritis Outcome Score) | 5 days postoperatively or until discharge
  According to physical examination by the orthopedics score KOOS (minimum 0, maximum 100) (higher score means better outcome)
Functionality of the prothesis - WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) | 5 days postoperatively or until discharge
  According to physical examination by the orthopedics score WOMAC (minimum 0, maximum 96) (higher score means worse outcome)
Functionality of the prothesis- G-FJS (German Forgotten Joint Score) | 5 days postoperatively or until discharge
  According to physical examination by the orthopedics score G-FJS (minimum 0, maximum 100) (higher score means better outcome)
Complications | 5 days postoperatively or until discharge
  Incidence of complications in total (e.g. delirium, allergic reactions, cardiopulmonary decompensation)
procedure specific time | during surgery
  time of the operation

CONTACTS AND LOCATIONS:
Overall Officials: Gregor A Schittek, MD, Principal Investigator — Med Uni Graz
Locations (1):
- Medical University Hospital LKH Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be made available upon reasonable request
Access Criteria: Data will be made available upon reasonable request